CLINICAL TRIAL: NCT02887430
Title: The Effect of Foot Reflexology Therapy on Pain Intensity and Health-related Quality of Life in People With Non-specific Low Back Pain
Brief Title: Foot Reflexology Therapy and Non-specific Low Back Pain
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universiti Sultan Zainal Abidin (Other)
Responsible Party: Principal Investigator, nor dalila marican, Principle investigator, Universiti Sultan Zainal Abidin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: UHREC/2016/2/011
Record Dates: First submitted 2016-08-19; First posted 2016-09-02 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Low Back Pain
Keywords: foot reflexology; pain intensity; health-related quality of life
MeSH Terms: conditions — Low Back Pain; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention (Experimental): Participants will be received 8 sessions of foot reflexology therapy, 30 minutes each (2 sessions per week of 4 weeks) and low back pain standard care
  Interventions: Other: foot reflexology therapy
- control (No Intervention): participants will be received standard care in general practice

INTERVENTIONS:
Other: foot reflexology therapy — standard care and foot reflexology
  Arms: intervention

SUMMARY:
The aim of this study was to investigate whether the eight therapy session with foot reflexology can reduce pain intensity when applied as an addition to the standards care of low back pain according to the Malaysian low back pain management guidelines.

DETAILED DESCRIPTION:
Low back pain is a common health complaint in most societies. Many treatments for low back pain aim to reduce suffering quicken recovery and minimize recurrence or development of chronic disability. However, low back pain continues as a societal enigma. The aim of this study was to investigate whether the eight therapy session with foot reflexology can reduce pain intensity when applied as an addition to standards care of low back pain according to the Malaysian low back pain management guidelines. Analysis of health-related quality of life will also be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Have been medically diagnosed with a non-specific low back pain.
* Have not received treatment for low back pain within the previous 2 weeks.
* Are at least 18 years old.
* Have both feet and all toes intact and free from wounds.
* Have not undergone any other complementary and alternative therapies during the study.

Exclusion Criteria:

* Have severe coexistent disease and serious pathology or systemic illness.
* Have a specific diagnosed cause of back pain (infection, tumour, osteoporosis, fracture, an inflammatory condition or cauda equine syndrome).
* Have plantar fasciitis.
* Lack the ability to read and write Malaysia language.
* Had plans to move out of the area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-09; Primary Completion 2016-10 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
mean time in days to the recovery of pain | 5 months
  the mean time in days to the recovery of pain is measured at the first day the patient scores 0 to 10 point on the visual analog scale (VAS)

SECONDARY OUTCOMES:
demographic information | 3 month
  demographic information including age, ethnicity, marital status, educational level, weight, height, household monthly income, smoking status, alcohol consumption, co-morbid disease and categories of low back pain.
side effects of treatment | 5 month
  reporting of possible side effects of the treatment, both reflexology and medication
health-related quality of life | 5 months
  measuring mean of health-related quality of life using Euro-quality of life 5D questionnaire before and after intervention

IPD SHARING:
Plan to Share IPD: Undecided